CLINICAL TRIAL: NCT05144659
Title: Evaluation of Double Faced Transverse Preputial Onlay Island Flap for Hypospadias Repair in Pediatrics.
Acronym: DFOF#TIOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Faculty of Medicine, Al-Azhar University, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Al-Azhar DFOF versus TIOF
Record Dates: First submitted 2021-11-20; First posted 2021-12-03 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Hypospadias
Keywords: Double face;; Onlay island flap;; Inner preputial flap;; Hypospadias in pediatrics
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Intervention Model Description: 68 pediatric patients will be randomly divided (using non-transparent closed envelope randomization method) into two equal groups, each will include 34 patients; Group A will undergo double-faced preputial onlay island flap and Group B will undergo transverse inner preputial onlay island flap.
Who Masked: Participant, Investigator
Masking Description: 2 (Participant, Investigator) 2 masking (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double faced transverse preputial onlay island flap (group A) (Active Comparator): Thirty-four patients undergo double faced transverse preputial onlay island flap are categorized as (group A)
  Interventions: Procedure: Double faced transverse preputial onlay island flap
- transverse inner preputial onlay island flap (control group) (group B) (Active Comparator): Another thirty-four patients undergo transverse inner preputial onlay island flap are categorized as the control group = (group B)
  Interventions: Procedure: Transverse inner preputial onlay island flap

INTERVENTIONS:
Procedure: Double faced transverse preputial onlay island flap — A well-established one-stage repair of penile hypospadias called Double faced transverse preputial onlay island flap
  Arms: Double faced transverse preputial onlay island flap (group A)
Procedure: Transverse inner preputial onlay island flap — A second well-established one-stage repair of penile hypospadias called Transverse inner preputial onlay island flap
  Arms: transverse inner preputial onlay island flap (control group) (group B)

SUMMARY:
Evaluation of double faced transverse preputial onlay island flap for hypospadias repair in pediatrics. The preputial onlay island flap technique has been popularized for hypospadias repair as a result of offering a consistent combination of excellent cosmetic results and acceptable complication rates. Like other techniques, urethrocutaneous fistulae continue to be the most common complications, in addition to other complications, and can be attributed to the affection of flaps vascularity. Some authors describe a technique that resolves some of these problems by combining the unique benefits of the double-faced preputial flaps.

This study aimed to evaluate double faced preputial onlay island flap technique for complication rate, outcomes for urinary stream, and cosmetic results.

DETAILED DESCRIPTION:
Type of study: prospective RCT

Review of literature:

* Different previous techniques for the repair of various levels of penile shaft hypospadias with chordee.
* Demonstration of two different well-established techniques for repair of anterior, mid-penile, and posterior penile hypospadias without or with mild curvature.
* Disadvantages of two-stage urethroplasty or technique as transverse inner preputial onlay island flap that involves dissection of the flap from its dorsal preputial tissue (as it affects the flap vascularity).
* Merits of single-stage urethroplasty double-faced preputial onlay island flap (as it combines the benefits of vascularized pedicled flap, provides better functional and cosmetic results, and low complication rate).

This study will be conducted at pediatric surgery department at Al-Houssain and Sayed Galal University Medical Centers, in the period from May 2019 to February 2021, on 68 male patients with anterior, mid-penile, and posterior penile hypospadias without or with mild curvature.

Patients will be investigated by routine laboratory tests for fitness for surgery. All of them will undergo one-stage repair using either of 2 techniques of urethroplasty; double-faced preputial onlay island flap versus transverse inner preputial onlay island flap.

Written informed consent will be signed by the parents of all participants in the study.

Institutes of the study: A multicenter study at pediatric surgery departments, Al-Azhar University Medical Centers in Cairo, Egypt.

Number of cases: Sixty-eight male patients. Time frame: 3 years.

Ethical Consideration:

The protocol will be discussed and approved by the Ethics and Institutional Review Board Committee at the investigators' hospitals. The procedures and the aim of the study will be clearly explained to the patient and the family. Written informed consent will be obtained before enrollment of the patients into the study. The family's refusal to give consent for one-stage repair is respected but does not deprive the patient of getting surgical care by two-stage repair.

Preoperative preparation:

All patients will be subjected to history taking, clinical examination, and necessary laboratory investigations (CBC, Coagulation profile, Urinalysis). Participants will receive a dose of single broad-spectrum antibiotic 30 min-1 hour before surgery.

Patients will be randomly divided (using non-transparent closed envelope randomization method) into two equal groups, each will include 34 patients; Group A will undergo double faced preputial onlay island flap and Group B will undergo transverse inner preputial onlay island flap. All operations were done by the same surgical team.

Follow-up: patients will be followed-up at OPD at 1, 3, 12, and 24 months, for incidence of any complications. HOSE score questionnaire will be used for the evaluation of outcomes.

Statistical Analysis:

Data will be presented as mean, standard deviation, number & percentage. For qualitative data, Chi-square test (X2) is used to compare between the two groups and independent-samples t-test of significance is used when comparing between two means. The significance level is set at P <0.05. Statistical analysis will be performed using statistical package for social sciences (SPSS) version 23.0, IBM Corp, IBM SPSS Statistics for Windows, Armonk, NY, USA.

Discussion:

It will focus on one-stage repair for anterior, mid-penile, and posterior penile hypospadias without or with mild penile curvature using double-faced preputial onlay island flap in comparison to inner preputial onlay island flap.

The results obtained from this study will be compared between both groups and with those reported in the literature.

Also, it will focus on results, complications, their management, and clinical evaluation by Hypospadias Objective Scoring Evaluation (HOSE) questionnaire evaluation tool. Finally, the investigators will conclude the reconstructive technique that gives the better results and least morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Young male pediatric patients diagnosed as anterior, mid-penile, or posterior penile hypospadias
* with shallow and narrow urethral plate measuring less than 6 millimeters,
* without or with mild penile curvature of less than 30º after degloving of the penis.

Exclusion Criteria:

* Patients with wide urethral plate suitable for tubularized incised plate (TIP) urethroplasty,
* other types of hypospadias as penoscrotal, scrotal, perineal hypospadias,
* patients with moderate or severe penile curvature,
* recurrent cases, and
* operations done by other surgeons

Ages: 1 Year to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male children with anterior, mid-penile, and posterior penile hypospadias without or with mild penile curvature
Enrollment: 68 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Urethrocutaneous fistula | 3 years
  Urethrocutaneous fistula in number of cases &percentage
Flap necrosis | 3 years
  Flap necrosis in number of cases &percentage
Glannular dehiscence | 3 years
  Glannular dehiscence in number of cases &percentage
Penile rotation | 3 years
  Penile rotation in number of cases &percentage
Urethral diverticulum | 3 years
  Urethral diverticulum in number of cases &percentage

SECONDARY OUTCOMES:
Meatal location | 3 years
  Meatal location in number of cases
Meatal shape | 3 years
  Meatal shape in number of cases
Urinary stream direction | 3 years
  Urinary stream in number of cases
Erection | 3 years
  Erection straightness in number of cases
Fistula | 3 years
  Fistula in number of cases

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abdelhaleem Hefney, MD, Study Chair — Pediatric Surgery Department, Al-Azhar University, Cairo, Egypt
Locations (1):
- Mohammad Alsayed Daboos, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be available for other researchers including methodology, figures, tables, results, and philosophy of discussion and the value this study will add to the literature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: November 2021 till indefinitely
Access Criteria: after the article became accepted and available online.
URL: http://orcid.org/0000-0002-6328-6419

REFERENCES:
- Available data/document: Study Protocol: orcid.org/0000-0002-6328-6419 — http://orcid.org/0000-0002-6328-6419 — Upon request of data, any researcher can e-mail the investigators at daboosmohammad@gmail.com or mohamedhafez_82@yahoo.com and the investigators will share the required data with the researchers and will be happy for any support.